CLINICAL TRIAL: NCT02616198
Title: A Prospective 6-year Clinical Study Evaluating Reinforced Glass Ionomer Cements With Resin Coating on Posterior Teeth
Brief Title: 6-year Clinical Evaluation of Glass Ionomer Cements (GIS) With Resin Coating on Posterior Teeth
Acronym: GIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sebnem Turkun, Prof. Dr., Ege University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-10.1/6
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Dental Caries
Keywords: glass ionomers; surface coating; clinical trial
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EquiaFil G-coat (Active Comparator): EquiaFil G-coat combination was applied on one randomly selected cavity to be restored
  Interventions: Other: EquiaFil Fuji Varnish; Other: Riva SC G-coat; Other: Riva SC Fuji Varnish
- EquiaFil Fuji Varnish (Active Comparator): EquiaFil Fuji Varnish combination was applied on one randomly selected cavity to be restored
  Interventions: Other: EquiaFil G-coat; Other: Riva SC G-coat; Other: Riva SC Fuji Varnish
- Riva SC G-coat (Active Comparator): River SC G-coat combination was applied on one randomly selected cavity to be restored
  Interventions: Other: EquiaFil G-coat; Other: EquiaFil Fuji Varnish; Other: Riva SC Fuji Varnish
- Riva SC Fuji Varnish (Active Comparator): River SC Fuji Varnish combination was applied on one randomly selected cavity to be restored
  Interventions: Other: EquiaFil G-coat; Other: EquiaFil Fuji Varnish; Other: Riva SC G-coat

INTERVENTIONS:
Other: EquiaFil G-coat — The old restorations or new caries were removed with anaesthetic solutions when necessary, a matrix was applied for two surface cavities and the restoration was performed with EquiaFil in bulk after mixing 10 sec. in the mixing machine. After 2min 30 sec, the restoration was contoured and the occlusion adjusted.Then the surface was coated with G-coat and light cured for 10 sec. The restorations were controlled by 2 independent examiners at baseline, 6-12-18 months and 6 years according to the United State Public Health Service criteria.
  Arms: EquiaFil Fuji Varnish; Riva SC Fuji Varnish; Riva SC G-coat
Other: EquiaFil Fuji Varnish — The old restorations or carious lesions were removed with anaesthetic solutions when necessary, a matrix was applied for two surface cavities and the restoration was performed with EquiaFil in bulk after mixing in the mixing machine. After 2min 30 sec, the restoration was contoured and the occlusion adjusted.Then the surface was coated in 2 layers of Fuji Varnish. The restorations were controlled by 2 independent examiners at baseline, 6-12-18 months and 6 years according to the United State Public Health Service criteria.
  Arms: EquiaFil G-coat; Riva SC Fuji Varnish; Riva SC G-coat
Other: Riva SC G-coat — The old restorations or carious lesions were removed and a sectional matrix was applied for two surface cavities and the restoration was performed with Riva SC in bulk after mixing 10 sec. in the mixing machine. The glass ionomer was packed with hand instruments in the cavities and 2min after the first setting the restoration was contoured and the occlusion adjusted.Then the surface was coated with G-coat resin and light cured for 10 sec. The restorations were controlled by 2 independent examiners at baseline, 6-12-18 months and 6 years according to the United State Public Health Service criteria.
  Arms: EquiaFil Fuji Varnish; EquiaFil G-coat; Riva SC Fuji Varnish
Other: Riva SC Fuji Varnish — The caries lesions were removed with diamond and stainless steel burs, a sectional matrix was applied for restoring two surface cavities and the restoration was performed with Riva SC in bulk after mixing 10 sec. in the mixing machine. After the first setting of 2min, the restoration was contoured and the occlusion adjusted.Then the surface was coated in 2 layers with Fuji Varnish. The restorations were controlled by 2 independent examiners at baseline, 6-12-18 months and 6 years according to the United State Public Health Service criteria.
  Arms: EquiaFil Fuji Varnish; EquiaFil G-coat; Riva SC G-coat

SUMMARY:
The aim of this study was to evaluate the long-term clinical performance of two highly viscous encapsulated GICs (EquiaFil and Riva SC) covered with two different coatings (Equia Coat and Fuji Varnish) over 6-year using modified United State Public Health Service (USPHS) criteria.

A total of 256 restorations were made with EquiaFil and Riva SC. Equia Coat or Fuji Varnish was used randomly on the surface of the restorations. The restorations were evaluated at baseline, 6, 12, 18 months and 6 years after placement using modified USPHS criteria. The results were evaluated with Pearson Chi-Square and Mann Whitney U-test (p< 0.05).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the long-term clinical performance of two highly viscous encapsulated GICs (EquiaFil and Riva SC) covered with two different coatings (Equia Coat and Fuji Varnish) over 6-year using modified United State Public Health Service (USPHS) criteria.

Fifty-four patients having Class I and II restorations/caries were included in the study. A total of 256 restorations were made with EquiaFil (GC Corp, Japan) and Riva SC (SDI, Australia). Equia Coat or Fuji Varnish was used randomly on the surface of the restorations. After cavity preparations, the teeth were randomly restored with one glass ionomer cement and coated with Equia Coat or Fuji Varnish. The restorations were evaluated at baseline, 6, 12, 18 months and 6 years after placement using modified USPHS criteria. Two evaluators checked color-match, marginal discoloration, marginal adaptation, caries formation, anatomical form, postoperative sensitivity and retention rate and photographs were taken at each recalls. The results were evaluated with Pearson Chi-Square and Mann Whitney U-test (p< 0.05).

The 18-month results were presented at the CED IADR congress iheld in Barcelona in 2010 (Turkun LS, & Kanic O ,Clinical evaluation of new glass ionomer coating combined systems for 18-months Journal of Dental Research 89 (Special Issue B) Abstract #402.) Gurgan S et al. also mentioned our 18-month results in their published manuscript ( Gurgan S,Kutuk ZB, Ergin E, Oztas ZZ & Cakir FY (2015) Four-year randomized clinical trial to evaluate the clinical performance of a glass ionomer restorative system Operative Dentistry 40(2) 134-143).

ELIGIBILITY:
Inclusion Criteria:

1. having good oral hygiene;
2. need for at least two or more posterior restorations in contact with neighbouring tooth and in occlusion with antagonist teeth;
3. teeth planned to be restore should be vital and symptomless;
4. the cavity isthmus size should be more than 1/3 of the intercuspal distance.

Exclusion Criteria:

1. absence of adjacent and antagonist teeth;
2. teeth with periodontal problems;
3. teeth with preoperative pain or pulpal inflammations;
4. teeth formerly subjected to direct pulp capping;
5. patients having severe systemic diseases, allergies or adverse medical history.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluating differently coated glass ionomer cements on posterior teeth with United State Public Health Service criteria regarding marginal adaptation by 2 independent evaluators | 6 years
  Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap (max 100µ) with discoloration (removable) Bravo: Marginal gap (> 100µ) with discoloration (unremovable) Charlie: The restoration is fractured or missed
Evaluating differently coated glass ionomer cements on posterior teeth with United State Public Health Service criteria regarding marginal discolouration by 2 independent evaluators | 6 years
  Marginal discolouration was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth.
  Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth.
  Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction.
Evaluating differently coated glass ionomer cements on posterior teeth with United State Public Health Service criteria regarding retention rate by 2 independent evaluators | 6 years
  Retention rate was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
Evaluating differently coated glass ionomer cements on posterior teeth with United State Public Health Service criteria regarding anatomic form by 2 independent evaluators | 6 years
  Anatomic form was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture
Evaluating differently coated glass ionomer cements on posterior teeth with United State Public Health Service criteria regarding colour changes by 2 independent evaluators | 6 years
  Colour changes was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed . A score means the higher score of clinical acceptability while C score means that the restoration has failed and needs to be replaced. Alpha: The restoration matches the adjacent tooth structure in color and translucency.
  Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth.
  Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency.

SECONDARY OUTCOMES:
Effects of resin coating on the performance of glass ionomer cements according to the United State Public Health Service criteria regarding marginal adaptation, marginal discolouration, retention rate, and colour changes by 2 independent evaluators | 6 years
  The effect of different coatings on the clinical performance of the different glass ionomers tested was evaluated with United State Public Health Service criteria at baseline, 6-12-18 months and 6-years. For the evaluation 2 independent evaluators using dental problem and mirrors evaluated the resin coatings according to their retention, marginal adaptation, marginal discolouration, and colour match. There were 4 evaluation scores. Alpha meaning a perfect resin coating, Bravo meaning a coating partially effective but still clinically acceptable and Charlie and Delta meaning that the coating was partially to totally missed.

REFERENCES:
- [Background] Sidhu SK. Glass-ionomer cement restorative materials: a sticky subject? Aust Dent J. 2011 Jun;56 Suppl 1:23-30. doi: 10.1111/j.1834-7819.2010.01293.x. PMID 21564113
- [Background] Lohbauer U (2010) Dental glass ionomer cements as permanent filling materials? Properties, limitations and future trends. Materials 3(1) 76-96.
- [Background] Diem VT, Tyas MJ, Ngo HC, Phuong LH, Khanh ND. The effect of a nano-filled resin coating on the 3-year clinical performance of a conventional high-viscosity glass-ionomer cement. Clin Oral Investig. 2014 Apr;18(3):753-9. doi: 10.1007/s00784-013-1026-z. Epub 2013 Jul 7. PMID 23832616
- [Background] Tyas MJ. Clinical evaluation of glass-ionomer cement restorations. J Appl Oral Sci. 2006;14 Suppl:10-3. doi: 10.1590/s1678-77572006000700003. PMID 19089080
- [Background] Frankenberger R, Garcia-Godoy F, Kramer N. Clinical Performance of Viscous Glass Ionomer Cement in Posterior Cavities over Two Years. Int J Dent. 2009;2009:781462. doi: 10.1155/2009/781462. Epub 2010 Feb 22. PMID 20339470
- [Background] Ersin NK, Candan U, Aykut A, Oncag O, Eronat C, Kose T. A clinical evaluation of resin-based composite and glass ionomer cement restorations placed in primary teeth using the ART approach: results at 24 months. J Am Dent Assoc. 2006 Nov;137(11):1529-36. doi: 10.14219/jada.archive.2006.0087. PMID 17082278
- [Background] Burke FJ, Siddons C, Cripps S, Bardha J, Crisp RJ, Dopheide B. Clinical performance of reinforced glass ionomer restorations placed in UK dental practices. Br Dent J. 2007 Jul 14;203(1):E2; discussion 40-1. doi: 10.1038/bdj.2007.529. Epub 2007 Jun 1. PMID 17546060
- [Background] Bonifacio CC, Werner A, Kleverlaan CJ. Coating glass-ionomer cements with a nanofilled resin. Acta Odontol Scand. 2012 Dec;70(6):471-7. doi: 10.3109/00016357.2011.639307. Epub 2011 Dec 12. PMID 22149968
- [Background] Friedl K, Hiller KA, Friedl KH. Clinical performance of a new glass ionomer based restoration system: a retrospective cohort study. Dent Mater. 2011 Oct;27(10):1031-7. doi: 10.1016/j.dental.2011.07.004. Epub 2011 Aug 15. PMID 21840585
- [Background] Basso M, Brambilla E, Benites MG, Giovannardi M & Ionescu AC (2015) Glass ionomer cement for permanent dental restorations: a 48-months, multi-center, prospective clinical trial Stomatology Education Journal 2(1) 25-35.
- [Background] Miletic I, Baraba A, Juic IB & Anic I (2013) Evaluation of a glass-ionomer based restoration system- a one year pilot study Journal of Minimum Intervention in Dentistry 6 87-95.
- [Background] Gurgan S, Kutuk ZB, Ergin E, Oztas SS, Cakir FY. Four-year randomized clinical trial to evaluate the clinical performance of a glass ionomer restorative system. Oper Dent. 2015 Mar-Apr;40(2):134-43. doi: 10.2341/13-239-C. Epub 2014 Oct 9. PMID 25299703